CLINICAL TRIAL: NCT07174817
Title: Weight Loss on IVF Outcomes in Overweight and Obese Infertile Women: a Randomized Controlled Trial
Brief Title: Weight Loss on IVF Outcomes in Overweight and Obese Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Fu Min, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018PHB114-01
Record Dates: First submitted 2025-07-05; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Infertility; Weight Loss; Obesity; IVF
MeSH Terms: conditions — Infertility; Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weight loss intervention (Experimental): The weight loss intervention group received dietary and exercise interventions for 3 months prior to the start of IVF, including: intake of low glycemic index (GI) foods; a daily net energy expenditure of 500-750 Kcal; adherence to a weekly schedule of moderate-intensity exercise 3-5 times. After 3 months, weight maintenance management continued in accordance with the patients' preferences.
  Interventions: Behavioral: weight loss
- control (No Intervention): The control group, with standard clinical care, managed their weight independently before undergoing IVF.

INTERVENTIONS:
Behavioral: weight loss — The weight loss intervention group underwent dietary and exercise programs for three months prior to initiating IVF treatment. These interventions included consuming foods with a low glycemic index (GI), achieving a daily net energy expenditure of 500-750 kcal, and engaging in moderate-intensity exercise 3-5 times per week. After the three-month period, weight maintenance was managed according to each patient's preferences.
  Arms: weight loss intervention

SUMMARY:
The aim of this study is to determine whether weight loss prior to in vitro fertilization (IVF) improves live birth outcomes in overweight and obese infertile women. The study prospectively analyzed 158 overweight and obese (BMI ≥ 24 kg/m2) infertile women, age between 20 and 36 years, undergoing their first assisted reproduction treatment at the Reproductive Center of Peking University People's Hospital from January 2019 to December 2020. They were randomly allocated to two groups: one for weight loss intervention(dietary and exercise management) for 3 months prior to IVF and the other for control. All patients underwent standard ovarian stimulation, oocyte retrieval, and embryo transfer according to the local reproductive center protocol. Statistical analyses included descriptive statistics, logistic regression, and ROC curve analysis

DETAILED DESCRIPTION:
Background: Elevated body mass index (BMI) is associated with poorer outcomes in infertile women undergoing assisted reproductive technology (ART). However, evidence for effective weight loss interventions and their impact on live birth rates remains limited and inconclusive. The aim of this study is to determine whether weight loss prior to in vitro fertilization (IVF) improves live birth outcomes in overweight and obese infertile women.

Methods: This randomized controlled clinical trial enrolled 158 overweight or obese (BMI ≥ 24 kg/m²) infertile women undergoing their first ART cycle at the Reproductive Center of Peking University People's Hospital. Participants were randomly allocated to either a weight intervention group or a control group using a computer-generated randomization sequence. The intervention group received a structured program consisting of dietary modification and physical exercise for three months prior to the initiation of IVF. In contrast, the control group received standard clinical care and were advised to manage their weight independently. The primary outcome measure was the live birth rate.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese infertile women attending the Reproductive Centre of Peking University People's Hospital for their first ART from January 2019 to December 2020

Exclusion Criteria:

* Women were excluded from enrolment if they had concomitant endocrine abnormalities, chromosomal abnormalities affecting pregnancy outcome, history of previous ovarian surgery, or malformed uterus.

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of participants with live birth | From Day 0 of the first embryo transfer cycle (cycle length: 28 days) through the entire pregnancy period until delivery, including both preterm and full-term births
  Live birth rate in overweight and obese infertile patients undergoing their first embryo transfer cycle, including premature and full-term birth

CONTACTS AND LOCATIONS:
Locations (1):
- Min Fu, Beijing, Beijing Municipality, China